CLINICAL TRIAL: NCT05016167
Title: The Effect of Replacement Frequency of Electrodes on Skin Moisture and Condition in Infants Hospitalized in the Pediatric Intensive Care Unit
Brief Title: The Effect of Replacement Frequency of Electrodes on Skin in Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assist. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2018/11
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Infant, Premature
Keywords: Infant; Moisture; Monitoring; Pediatric Intensive Care; Skin
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (replacement every 24 hours) (Other): The monitoring electrodes were not replaced for 24 hours, the electrodes were removed at the end of 24 hours (the protocol currently used in the institution) in control group.
  Interventions: Procedure: Replacement every 24 hours
- Experimental Group (replacement every 12 hours) (Experimental): In the experimental group, the monitoring electrodes were replacement every 12 hours within 24 hours.
  Interventions: Procedure: Replacement every 12 hours

INTERVENTIONS:
Procedure: Replacement every 24 hours — Processing Steps:
  1. The monitoring electrodes were not replaced for 24 hours, the electrodes were removed at the end of 24 hours. During the 24-hour follow-up, patients whose electrodes were removed for any reason were excluded from the sample.
  2. Immediately after the drying, skin moisture measurement was made in the right 2nd intercostal space (ICA), left 2nd ICA, and midclavicular 5th ICA regions.
  3. The skin condition was evaluated from the areas monitored using the skin condition score by the researcher and another independent observer.
  4. The data were recorded.
  Arms: Control group (replacement every 24 hours)
Procedure: Replacement every 12 hours — Processing Steps:
  1. Monitoring electrodes were removed at the end of the 12th hour. When removing the monitoring electrodes, the area was first wetted using a disinfectant and dried using a sponge after removing the electrodes.
  2. Immediately after the drying, skin moisture measurement was made in the right 2nd ICA, left 2nd ICA and midclavicular 5th ICA regions.
  3. The skin condition was evaluated from these areas monitored using the skin condition score by the researcher and another independent observer.
  4. Monitored again.
  5. Monitoring electrodes were removed at the end of the 24th hour. Cleaning and drying were done immediately after removal.
  6. Immediately after drying, skin moisture was measured from the monitored areas.
  7. The skin condition was evaluated from the areas monitored using the skin condition score by the researcher and another independent observer.
  8. The data were recorded.
  Arms: Experimental Group (replacement every 12 hours)

SUMMARY:
In the Pediatric Intensive Care Unit (PICU), each child and infant is monitored to determine the status of the underlying disease by constantly monitoring the main variables, to help diagnosis and to guide treatment. During the monitoring application, electrodes of appropriate size for the patient's age and body surface are attached to the appropriate areas of the patient where skin integrity is intact, clean, and dry. It is recommended that these electrodes be replaced within 24 hours at most, but there is no evidence of the effect of electrode replacement frequency on skin moisture and integrity.

Based on this reason, this study was conducted experimentally in a randomized controlled manner to determine the effect of frequency of monitoring electrode replacement on skin moisture and condition of infants hospitalized in the PICU.

DETAILED DESCRIPTION:
The study was conducted with 66 participants, with the number of participants being 33 in both two groups (Experimental and Control Group).The randomization of the sample was determined by entering the total number of cases in line with the Research Randomizer program.

The control group of the study involved infants whose monitoring electrodes were replaced at the 24th hour after being monitored and the experimental group involved infants whose monitoring electrodes were replaced at the 12th and 24th hour after being monitored.

Before all participants are monitored, skin cleansing was performed on the right second intercostal space (Right 2nd ICA), left second intercostal space (Left 2nd ICA) and the left lower side of the sternum at the left midclavicular level in the fifth intercostal space (Midclavicular 5th ICA). After that, skin moisture was measured where monitoring will be performed and skin condition evaluation of these areas. Then the participants were monitored.

After these applications, skin moisture and skin condition score evaluations were repeated in both groups.

Skin Condition Score The skin condition score, developed by the Association of Women's Health, Obstetric and Neonatal Nurses (AWHONN) and validated by Calisir et al. in 2016, was used to determine the skin condition. The scale consists of three items and each item includes an evaluation criterion. These are dryness, erythema, and skin integrity breakdown/peeling, respectively. Each item of the 3-point Likert scale gets 1 to 3 points. The lowest score that can be obtained from the scale is 3, the highest score is 9. A high total score indicates that the skin condition of the newborn is poor. Permission was obtained for the use of the skin condition score from the Association of Women's Health, Obstetric and Neonatal Nurses (AWHONN) and the authors who performed the Turkish validity and reliability.

Skin Moisture Digital Moisture Monitor For Skin was used to measure skin moisture. This moisture measuring device measures with "%". This device developed for precise measurement has been preferred because of its ability to show the amount of moisture by the contact without damaging the skin, being portable, working with a battery, having a wide measurement range (it can measure the amount of skin moisture from 0% to 99.9%), because of its fast, easy and reliable use, low cost, and its ability to measure in many anatomical regions.

Materials provided in accordance with the procurement procedure of the institution where the research was conducted and used in patient care during the data collection phase were preferred as consumable materials.

Researchers do not have any conflict of interest with companies regarding the preference of these materials. The consumables that are still used in the institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose parents agreed to participate in the study and signed the informed consent form
* No history of surgical procedures
* Recently admitted to the unit and monitored for the first time
* Infants aged ≥ 1 to 12 ≤ months

Exclusion Criteria:

* Infants with a skin disease, with other diseases that can affect skin moisture and condition, with immune system disease

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Change in skin moisture | Data collected immediately before monitoring, after monitoring 12th hour (only for experimental group) and after 24 th hours. The change in these time intervals assessed.
  Digital Moisture Monitor For Skin was used to measure skin moisture. This moisture measuring device measures with "%". This device developed for precise measurement has been preferred because of its ability to show the amount of moisture by the contact without damaging the skin, being portable, working with a battery, having a wide measurement range (it can measure the amount of skin moisture from 0% to 99.9%). As the moisture in the skin increases, the % increases.
  Skin moisture measurement was made in the right 2nd ICA, left 2nd ICA, and midclavicular 5th ICA regions.
Change in skin condition | Data collected immediately before monitoring, after monitoring 12th hour (only for experimental group) and after 24 th hours. The change in these time intervals assessed.
  Skin condition were evaluated with the Skin Condition Assessment Scale. The scale consists of three items and each item includes an evaluation criterion. These are dryness, erythema, and skin integrity breakdown/peeling, respectively. Each item of the 3-point Likert scale gets 1 to 3 points. The lowest score that can be obtained from the scale is 3, the highest score is 9. A high total score indicates that the skin condition of the newborn is poor.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Onturk, Assist Prof, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University Atakent Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flodgren G, Conterno LO, Mayhew A, Omar O, Pereira CR, Shepperd S. Interventions to improve professional adherence to guidelines for prevention of device-related infections. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD006559. doi: 10.1002/14651858.CD006559.pub2. PMID 23543545
- [Result] Gray M, Black JM, Baharestani MM, Bliss DZ, Colwell JC, Goldberg M, Kennedy-Evans KL, Logan S, Ratliff CR. Moisture-associated skin damage: overview and pathophysiology. J Wound Ostomy Continence Nurs. 2011 May-Jun;38(3):233-41. doi: 10.1097/WON.0b013e318215f798. PMID 21490547
- [Result] Voegeli D. Prevention and management of moisture-associated skin damage. Nurs Stand. 2019 Jan 25;34(2):77-82. doi: 10.7748/ns.2019.e11314. PMID 31468844
- [Result] Delmore B, Deppisch M, Sylvia C, Luna-Anderson C, Nie AM. Pressure Injuries in the Pediatric Population: A National Pressure Ulcer Advisory Panel White Paper. Adv Skin Wound Care. 2019 Sep;32(9):394-408. doi: 10.1097/01.ASW.0000577124.58253.66. PMID 31436620
- [Result] Widiati E, Nurhaeni N, Gayatri D. Medical-Device Related Pressure Injuries to Children in the Intensive Care Unit. Compr Child Adolesc Nurs. 2017;40(sup1):69-77. doi: 10.1080/24694193.2017.1386973. PMID 29166186
- [Result] Jackson D, Sarki AM, Betteridge R, Brooke J. Medical device-related pressure ulcers: A systematic review and meta-analysis. Int J Nurs Stud. 2019 Apr;92:109-120. doi: 10.1016/j.ijnurstu.2019.02.006. Epub 2019 Feb 10. PMID 30782513
- [Derived] Demirci K, Ugur E, Onturk ZK. Replacing Monitoring Electrodes on Infant Skin Every 12 Versus 24 Hours. Adv Skin Wound Care. 2023 Aug 1;36(8):1-8. doi: 10.1097/ASW.0000000000000010. PMID 37471452